CLINICAL TRIAL: NCT06290427
Title: Comparison of Outcomes of Multiple Platforms for Assisted Robotic-Kidney
Brief Title: Comparison of Outcomes of Multiple Platforms for Assisted Robotic-Kidney (COMPAR-K)
Acronym: COMPAR-K
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Alessandro Antonelli, MD, Prof, MD, Director of Urology Unit, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: COMPAR-K
Record Dates: First submitted 2024-02-21; First posted 2024-03-04 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Renal Carcinoma
Keywords: Robotic-assisted surgery; Partial Nephrectomy; Multiple surgical platforms; Postoperative complications; Operative outcomes
MeSH Terms: conditions — Carcinoma, Renal Cell; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- DaVinci system (Active Comparator): Robot-assisted partial nephrectomy is performed using the DaVinci platform
  Interventions: Device: DaVinci RAPN
- Hugo RAS system (Experimental): Robot-assisted partial nephrectomy is performed using the Hugo RAS platform
  Interventions: Device: Hugo RAS RAPN

INTERVENTIONS:
Device: DaVinci RAPN — Robot-assisted Partial Nephrectomy with DaVinci® Surgical System
  Arms: DaVinci system
Device: Hugo RAS RAPN — Robot-assisted Partial Nephrectomy with Hugo™ RAS System
  Arms: Hugo RAS system

SUMMARY:
The Urology Unit of AOUI Verona proposes a clinical study aimed at a preliminary evaluation of postoperative complications specifically focused on robotic partial nephrectomy (RAPN) procedures using two currently available platforms:

* DaVinci®;
* Hugo®.

The questions it aims to answer are:

Does the estimation of the post-operative complications suggest something? Are differences (intra- and post-operative, oncological, functional, technical, and economic) among the three intervention approaches observable?

Participants will be invited to join one of these two experimental group:

1. surgery with the DaVinci platform;
2. surgery with the Hugo platform.

ELIGIBILITY:
Inclusion Criteria:

* patient aged between 18 and 90 years old;
* patient with localized kidney tumor suitable for partial nephrectomy;
* patient able to understand and sign the informed consent;
* patient compliance with the follow-up program.

Exclusion Criteria:

* patient who do not fall within the inclusion age range;
* patient not suitable for partial nephrectomy;
* patient unable to understand and sign the informed consent;
* patient unable to follow the monitoring program;
* patient refusal to participate to the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with postoperative complications | Over the 4 days post surgery
  Overall postoperative complications (% score >0) are considered by Clavien-Dindo Classification 7 grades (I, II, IIIa, IIIb, IVa, IVb and V): the higher the grade, the higher the severity of the complication
Number of participants with moderate to major postoperative complications | Over the 4 days post surgery
  Moderate to major complications (% score >=2) are considered by Clavien-Dindo Classification 7 grades (I, II, IIIa, IIIb, IVa, IVb and V): the higher the grade, the higher the severity of the complication
Number of participants with major postoperative complications | Over the 4 days post surgery
  Major complications (% score >=3) are considered by Clavien-Dindo Classification 7 grades (I, II, IIIa, IIIb, IVa, IVb and V): the higher the grade, the higher the severity of the complication

SECONDARY OUTCOMES:
Overall duration of the surgery | Intraoperative
  Minutes
Number of intraoperative complications | Intraoperative
  Proportion of events
Type of intraoperative complications | Intraoperative
  Note of the event detail
Number of intraoperative technical malfunctions | Intraoperative
  Proportion of events
Type of intraoperative technical malfunctions | Intraoperative
  Note of the event detail
Estimated Blood Loss | Intraoperative
  Volume
Postoperative hospitalization | From the day after surgery up to 10 days postoperative
  Days of recovery until the date of discharge
Postoperative pain | 1-4 days postoperative
  Numerical Rating Scale (NRS) 0-10 scale for the self-reported rate of pain: zero meaning "no pain" and 10 meaning "the worst pain imaginable"
Positive Surgical Margins | Up to 2 weeks postoperative (at the end of histological analysis)
  Rate after histological examination
Serum Creatinine dosage for renal function assessment | 1 month, 3 and 6 months follow-up
  Creatinine test
Estimated Glomerular Filtration Rate for renal function assessment | 1 month, 3 and 6 months follow-up
  eGFR calculation estimated by EPI-CKD formula
Time taken for platform related timings | From the room setting, through the overall surgical procedure, until postoperative room restoration for each of expected 45 surgeries (through study completion: about 4 months)
  Configuration of the surgical table, Draping, Undraping, Docking, Undocking
Procedure-related costs | From surgical procedure to the end of follow-up period (6 months)
  Estimate

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro AA Antonelli, MD, Principal Investigator — Azienda Ospedaliera Universitaria Integrata Verona
Locations (1):
- Urology Unit, AOUI Verona, Verona, VR, Italy